CLINICAL TRIAL: NCT00437970
Title: Drug naïve Indigenous Australians With Type 2 Diabetes, Enrolled in a Randomised Controlled Trial of Rosiglitazone Versus Metformin Monotherapy to Assess the Effects on Metabolic and Cardiovascular Parameters
Brief Title: Medication in Early Diabetes (MED) Study
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to secure supply of the study medication
Sponsor: Menzies School of Health Research (Other)
Responsible Party: The Director, Menzies School of Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DART-MSHR-06-29
Record Dates: First submitted 2007-02-18; First posted 2007-02-21 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Arm A- Metformin
  Interventions: Drug: Metformin
- B (Active Comparator): Arm B- Pioglitazone
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — 15mg of Pioglitazone taken orally twice a day
  Arms: B
Drug: Metformin — 500 mg of Metformin taken orally twice a day
  Arms: A

SUMMARY:
This study compares metformin (current first-line medication) to pioglitazone (a newer diabetic medication currently approved for combination use). Whilst there is good evidence for the benefits of pioglitazone use in other populations, in light of the known weight gain effects of pioglitazone we believe further assessment is required in Indigenous Australians (in whom there is a strong predisposition for central fat deposition). This study will provide evidence regarding the medication appropriate for first line medication in Type 2 diabetes in this high risk population. This study will assist clinicians to make evidenced-based decisions regarding initial medical management of those with Type 2 diabetes (where there is currently a gap in evidence).

ELIGIBILITY:
Inclusion Criteria:

* Drug naïve Indigenous Australians with Type 2 Diabetes
* Permanent resident of Darwin for at least 1 year immediately before and expected to be for at least 1 year after study commences
* Participants must be able to give informed voluntary consent
* Both males and females (females of child bearing potential excluded if not on reliable means of contraception)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
HbA1c values | second monthly
Weight gain | monthly
Weight distribution | six monthly
Medication side effects | monthly

SECONDARY OUTCOMES:
Medication compliance | monthly
Side effects | monthly
Lipids | second monthly
Endothelial dysfunction. | second monthly

CONTACTS AND LOCATIONS:
Overall Officials: Louise Maple Brown, MBBS PhD FRACP, Principal Investigator — Menzies School of Health Research
Locations (1):
- Menzies School of Health Research, Darwin, Northern Territory, Australia

REFERENCES:
- See also: Related Info — http://www.menzies.edu.au